CLINICAL TRIAL: NCT00580658
Title: Humanitarian Device Exemption for Medtronic Activa Dystonia Therapy
Brief Title: Humanitarian Device Exemption
Acronym: Dystonia IRB
Status: Approved for marketing | Type: Expanded Access
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Peter Konrad, Professor, Director of Functional Neurosurgery, Vanderbilt University
Other Study IDs: 060155
Record Dates: First submitted 2007-12-13; First posted 2007-12-27 (Estimated); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Dystonia
Keywords: Dystonia; DBS
MeSH Terms: conditions — Dystonia

INTERVENTIONS:
Device: Medtronic Activa Gpi — Activa Therapy, Gpi
  Other Names: DBS; Gpi; Activa Therapy

SUMMARY:
The purpose of this study is to allow patients to undergo deep brain stimulation (DBS) surgery for the treatment of dystonia. This is NOT a research study, but rather, a requirement by the FDA for humanitarian use of the deep brain stimulator device in the treatment of this rare disorder. Use of DBS for dystonia is approved for humanitarian use by the FDA in the treatment of chronic, intractable (drug refractory) dystonia, including generalized and segmental dystonia, hemidystonia, and cervical dystonia (torticollis) in patients 7 years or older. Thus, this proposal request authorization by the IRB to allow patients at VUMC to access this HUD therapy.

DETAILED DESCRIPTION:
The purpose of this IRB approved study is to allow patients to undergo deep brain stimulation (DBS) surgery for the treatment of dystonia. This is NOT a research study, but rather, a requirement by the FDA for humanitarian use of the deep brain stimulator device in the treatment of this rare disorder. Use of DBS for dystonia is approved for humanitarian use by the FDA in the treatment of chronic, intractable (drug refractory) dystonia, including generalized and segmental dystonia, hemidystonia, and cervical dystonia (torticollis) in patients 7 years or older. Thus, this proposal request authorization by the IRB to allow patients at VUMC to access this HUD therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose ages are in the range of 7 and 99 years old
* Patients who are diagnosed with chronic, intractable (drug refractory)primary dystonia, including generalized and or segmental dystonia, hemidystonia, and cervical dystonia (torticollis)as determined by a neurologist or neurosurgeon.
* Patients who have failed appropriate medical therapy as determined by the SMD conference

Exclusion Criteria:

* Patients younger than 7 years old
* Patients who are at significant surgical risk as determined by the neurosurgeon and/or anesthesiologist.
* Patients who have not had an adequate trial of medical or non-surgical therapy as determined by the SMD conference.
* Patients not deemed good candidates by the SMD conference group.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Peter E Konrad, MD, Ph.D., Principal Investigator — Vanderbilt University, Dept. Neurosurgery; Dario Englot, MD PhD, Principal Investigator — Vanderbilt University, Dept. Neurosurgery; Thomas L Davis, MD, Principal Investigator — Vanderbilt University, Dept. Neurology; John Y Fang, MD, Principal Investigator — Vanderbilt University, Dept. Neurology
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States